CLINICAL TRIAL: NCT02241447
Title: Study to Improve Outcomes in Aortic Stenosis. International, Multi-center, Prospective, Observation and Interventional Cohort Registry
Brief Title: Quality of Care in AS IMPULSE Study
Acronym: IMPULSE
Status: Completed | Type: Observational
Sponsor: Institut für Pharmakologie und Präventive Medizin (Network)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: IMPULSE
Record Dates: First submitted 2014-09-02; First posted 2014-09-16 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Aortic Valve Stenosis
Keywords: aortic valve Stenosis; Echo; TAVI; SAVR; referral
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Observation: the nurse identifies cases with severe AS and collects their data. Baseline data for each patient will be collected and a follow-up will be done after three months for each patient to determine his/her outcome and the treatment that was decided on
- Early information: in this arm, the physician referring a patient for echocardiography will be notified of a finding of severe aortic stenosis: the nurse brings cases with severe AS to the attention of the referring physician within a week (via phone, e-mail or letter) to make them aware of the diagnosis.

SUMMARY:
The purpose of this study is to narrow the gap between patients being diagnosed with severe aortic stenosis and those being appropriately monitored and treated. For this purpose a prospective survey of current practice (3 months) will be conducted followed by a six month period of intervention during which a variety of quality improvements measures will be implemented. There will then be a 3 month follow-up period during which the legacy of this initiative will be monitored during which no intervention will be carried out.

DETAILED DESCRIPTION:
All patients meeting pre-specified criteria (severe aortic stenosis whether with or without symptoms) will be collected. There will be three phases at each site observation A, intervention, observation B. Observation A: In this phase, the nurse identifies cases with severe AS and collects their data. Baseline data for each patient will be collected and a follow-up will be done after three months for each patient to determine his/her outcome and the treatment that was decided on. There will also be an optional telephone follow-up to find out the patient's outcome.

Intervention: In this phase, the physician referring a patient for echocardiography will be notified of a finding of severe aortic stenosis: the nurse brings cases with severe AS to the attention of the referring physician within a week (via phone, e-mail or letter) to make them aware of the diagnosis.

Baseline and follow-up data will be collected for each patient as before. Moreover, more detailed data with regard to the patient's health status will be documented.

Observation B: Same as Observation Phase A

ELIGIBILITY:
Inclusion Criteria:

* Aortic valve area < 1cm2
* Indexed aortic valve area <0.6 cm/m2
* Maximum Jet velocity > 4.0 m/sec
* Mean transvalvular gradient > 40 mmHg

Exclusion Criteria:

* Non-severe aortic Stenosis (AS)
* Previous aortic valve replacement (AVR)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged over 18years identified on echocardiography with severe AS
Sampling Method: Non-Probability Sample
Enrollment: 2173 (Actual)
Dates: Start 2014-08-08 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Referral rates at 3 months for Intervention (SAVR or TAVI) | 3 months

SECONDARY OUTCOMES:
Referral rates at 3 months for exercise testing or stress echocardiography | 3 months
Time to next out-patient appointment or clinical review | 15 months
Type of intervention selected (SAVR, TAVI, watchful waiting or no treatment) | 3 months
Appropriateness of treatment decisions made in collaboration with the valve specialist | 3 months
Outcomes (survival) at 1 year (telephone FU) including the time between diagnosis and treatment | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard Steeds, MD, Principal Investigator — Queen Elizabeth Hospital, Birmingham, UK; Norbert Frey, MD, Principal Investigator — Department of Cardiology and Angiology, University of Kiel, Germany; Davia Messika-Zeitoun, MD, Principal Investigator — Hôpital Bichat, Paris FR
Locations (23):
- Krankenhaus Hietzing, Vienna, Austria
- IKEM - Institute for Clinical and Experimental Medicine, Prague, Czechia
- France (2):
  - Centre Hospitalier d'Annecy, Annecy
  - Bichat Hospital, Paris
- Germany (8):
  - Charité - Campus Benjamin Franklin, Berlin
  - Herzzentrum Universitätsklinikum Köln, Cologne
  - Universitätsklinikum Erlangen, Erlangen
  - Westpfalz Klinikum, Kaiserslautern
  - UKSK Campus Kiel, Klinik für Kardiologie und Angiologie, Kiel
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Städtisches Klinikum München, München
  - Krankenhaus der Barmherzigen Brüder, Trier
- Italy (5):
  - Università degli Studi di Bari Aldo Moro, Bari
  - University "Magna Græcia" of Catanzaro, Catanzaro
  - IRCCS San Matteo Hospital, Pavia
  - Policlinico Umberto I Rom, Rome
  - University of Torino, Torino
- AMC Medical Center, Amsterdam, Netherlands
- Santa Creu Barcelona, Barcelona, Spain
- UniversitätsSpital Zürich, Zurich, Switzerland
- United Kingdom (3):
  - Queen Elizabeth Hospital, Birmingham
  - Bart Heart Center, London
  - James Cook University Hospital, Middlesbrough

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Steeds RP, Lutz M, Thambyrajah J, Serra A, Schulz E, Maly J, Aiello M, Rudolph TK, Lloyd G, Bortone AS, Hauptmann KE, Clerici A, Delle-Karth G, Rieber J, Indolfi C, Mancone M, Belle L, Lauten A, Arnold M, Bouma BJ, Deutsch C, Kurucova J, Thoenes M, Bramlage P, Frey N, Messika-Zeitoun D. Facilitated Data Relay and Effects on Treatment of Severe Aortic Stenosis in Europe. J Am Heart Assoc. 2019 Oct;8(19):e013160. doi: 10.1161/JAHA.119.013160. Epub 2019 Sep 24. PMID 31549578
- [Derived] Frey N, Steeds RP, Rudolph TK, Thambyrajah J, Serra A, Schulz E, Maly J, Aiello M, Lloyd G, Bortone AS, Hauptmann KE, Clerici A, Delle Karth G, Rieber J, Indorfi C, Mancone M, Belle L, Lauten A, Arnold M, Bouma BJ, Lutz M, Pohlmann C, Kurucova J, Thoenes M, Bramlage P, Messika-Zeitoun D; IMPULSE registry group. Symptoms, disease severity and treatment of adults with a new diagnosis of severe aortic stenosis. Heart. 2019 Nov;105(22):1709-1716. doi: 10.1136/heartjnl-2019-314940. Epub 2019 Jul 13. PMID 31302639
- See also: Related Info — https://europepmc.org/article/PMC/6806053
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/31302639